CLINICAL TRIAL: NCT05183412
Title: Effect of Virtual Reality (VR) Therapy on Patients Undergoing Hand Surgery Under Ultrasound-guided Regional Anesthesia: a Randomized Controlled Superiority Trial.
Brief Title: Effect of Virtual Reality (VR) Therapy on Patients Undergoing Hand Surgery Under Ultrasound-guided Regional Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principle Investigator, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: f/2021/126
Record Dates: First submitted 2022-01-05; First posted 2022-01-10 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Anesthesia, Local; Surgery; Hand Injuries
Keywords: Virtual reality glasses; Heart rate variability
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two independent assessors will gather data in this study: one blinded and one unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-guided regional nerve block and hand surgery without VR glasses (Active Comparator): Patients will not receive the VR glasses during the ultrasound-guided regional nerve block (axillary or distal peripheral) and hand surgery.
  Interventions: Procedure: Ultrasound-guided regional nerve block and hand surgery without VR glasses
- Ultrasound-guided regional nerve block and hand surgery with VR glasses (Experimental): Patients will receive the VR glasses during the ultrasound-guided regional nerve block (axillary or distal peripheral) and hand surgery.
  Interventions: Device: The Sedakit Oncomfort VR glasses (30-minutes Aqua program); Procedure: Ultrasound-guided regional nerve block and hand surgery with VR glasses

INTERVENTIONS:
Device: The Sedakit Oncomfort VR glasses (30-minutes Aqua program) — During placement of ultrasound-guided regional nerve block (axillary or distal peripheral) and hand surgery, patients are subjected to a 30-minutes VR program (Oncomfort SA, Wavre, Belgium) 'Aqua' via a head-mounted display and headphone. The patients watch a VR underwater view of the ocean while listening to speeches to induce relaxation and meditation.
  Arms: Ultrasound-guided regional nerve block and hand surgery with VR glasses
Procedure: Ultrasound-guided regional nerve block and hand surgery without VR glasses — During placement of ultrasound-guided regional nerve block (axillary or distal peripheral) and hand surgery, patients are NOT subjected to a 30-minutes VR program (Oncomfort SA, Wavre, Belgium) 'Aqua' via a head-mounted display and headphone.
  Arms: Ultrasound-guided regional nerve block and hand surgery without VR glasses
Procedure: Ultrasound-guided regional nerve block and hand surgery with VR glasses — Ultrasound-guided regional nerve block and hand surgery with VR glasses
  Arms: Ultrasound-guided regional nerve block and hand surgery with VR glasses

SUMMARY:
By means of an investigator-initiated, monocentric, single-blinded, prospective, randomized controlled superiority trial, the effect of virtual reality (VR) therapy on patients undergoing ambulatory hand surgery under ultrasound-guided regional nerve block will be investigated. It is hypothesized that the usage of VR during the placement of the nerve block in ambulatory hand surgery patients provides a significant decrease in pain score during anesthesia compared to without VR glasses. Additionally, an objective stress related parameter (HRV), anxiety, VR experience (immersion and presence), adverse effects and patient satisfaction are evaluated before anesthesia, during anesthesia and surgery or after surgery through validated questionnaires or measurements.

DETAILED DESCRIPTION:
Ultrasound-guided regional anesthesia (RA) is the golden standard in ambulatory superficial hand surgery due to its safety and reliability. Frequently used RA techniques are ultrasound-guided distal peripheral nerve block of the n. medianus and n. ulnaris is and ultrasound-guided axillary nerve block of the n. medianus, n. ulnaris, n. radialis, and n. musculocutaneous. The needling is frequently accompanied by stress, fear or anxiety and it has been proven in studies that psychological factors can affect the sensation of pain. At this moment systemic opioids and/or sedatives used, however, these partially neutralize the benefits of locoregional techniques.

Virtual reality (VR) is a non-pharmacologic and non-invasive simulation in which the user can interact within a 3D-computer-generated environment using special glasses with a screen and a headset. VR offers the ability to distract patients from reality and can therefore relieve a pain sensation from harmful stimuli. An important aspect of pain reduction in VR is presence and immersion. The physical/sensory stimulus offered by the artificial environment is referred to as immersion. Presence can be defined as one's sense of being in an artificial environment. The VR glasses of the firm Oncomfort called Sedakit™ have been proven to be safe and effective in previous clinical trials. A VR program namely 'Aqua', has been provided and designed for relaxation and distraction from anxiety or pain of patients.

Current literature is lacking objective parameters of stress within an operative, anesthesiologic framework. One of these objective stress-related parameters of is heart rate variability (HRV). HRV is the fluctuation of the length between consecutive heart beats and refers to the heart's ability to react to a wide range of physiological and environmental stimuli such as stress. HRV can be measured by the Empatica E4 wristband.

The proposed study, performed at the Jessa hospital, will assess the effect of VR glasses on pain levels of hand surgery patients during placement of the nerve block and surgery by comparing a group with VR glasses to without VR glasses. It is hypothesized that the usage of VR during the placement of the nerve block in ambulatory hand surgery patients provides a significant decrease in pain score during anesthesia compared to without VR glasses. Additionally, an objective stress related parameter (HRV), anxiety, VR experience (immersion and presence), adverse effects and patient satisfaction are evaluated before anesthesia, during anesthesia and surgery or after surgery through validated questionnaires or measurements.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years and <65 years
* ASA (American Society of Anesthesiology) classification: 1 - 3
* Patient scheduled for ambulatory hand surgery using ultrasound-guided axillary block regional anesthesia or ultrasound-guided peripheral nerve block.

Exclusion Criteria:

* Bilateral surgery
* BMI ≥ 40 kg/m²
* Motion sickness
* Patient that take medication that affects heart rhythm (beta-blockade)
* Infection in the area for peripheral nerve block injections.
* Existing neurological conditions.
* Chronic pain symptoms
* Opioid use within the past 3 months
* Allergy to local anesthetics
* Inability to experience the VR glasses experience (Vision disorders)
* Inability to understand study design or mental impairment
* Patients with autonomic nervous system dysfunction
* Pregnancy
* Heart transplant patients, patients with diabetic neuropathy, patients with myocardial infarction (or having passed through it) and/or tetraplegic patients
* Fear of being under water
* Sea sickness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Pain due to the placement of the ultrasound-guided regional anesthesia block: Numeric Rating Scale (NRS) | Procedure (At the end of performing the ultrasound-guided regional anesthesia block)
  Pain caused by performing the anesthesia technique (measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)

SECONDARY OUTCOMES:
Pain due to the surgery: Numeric Rating Scale (NRS) | Intraoperative (At the end of surgery)
  Pain caused by performing the hand surgery (measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)
Stress: Heart rate variability (HRV) | Before performing the ultrasound-guided regional anesthesia block for 5 minutes in rest (baseline), procedure (during performing the ultrasound-guided regional anesthesia block ) and minute 0 - 5 during the surgical procedure.
  Heart rate variability (HRV), is the fluctuation of the length between consecutive heart beats in milliseconds and is regulated by the autonomic nerve system. It determines the balance between the parasympathetic 'rest and digest' and sympathetic 'flight or fight' nerve systems. The sympathetic branch decreases HRV during stressful situations, while the parasympathetic branch increases HRV at rest. This natural interplay between the two systems allows the heart to quickly respond to different stimuli, including stress. HRV (being RMSSD and HF-HRV), is measured during placement of an ultrasound-guided regional anesthesia block and surgery through the Empatica E4 wristband (Photoplethysmography).
Anxiety due to placement of the ultrasound-guided regional anesthesia block: Numeric Rating Scale (NRS) | Procedure (At the end of performing the ultrasound-guided regional anesthesia block)
  Anxiety caused by performing the anesthesia technique (measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)
Anxiety due to the surgery: Numeric Rating Scale (NRS): Numeric Rating Scale (NRS) | Intraoperative (At the end of surgery)
  Anxiety caused by performing the hand surgery (measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)
Pre-surgical anxiety (Surgical Fear Questionnaire) | Arrival at the 1 day clinic
  Pre-surgical anxiety for the anesthesia and surgery (measured with the Surgical Fear Questionnaire)
VR experience: Immersion and presence (Igroup questionnaire) | Intraoperative (At the end of surgery)
  An important aspect of pain reduction in VR is presence and immersion. The physical/sensory stimulus offered by the artificial environment is referred to as immersion. Presence can be defined as one's sense of being in an artificial environment.
Adverse effects (Simulation Sickness Questionnaire and Virtual Reality Symptom Questionnaire) | Intraoperative (At the end of surgery)
  Adverse effects (dizziness, headache, motion sickness, postoperative nausea and vomiting, fatigue, claustrophobia) are evaluated by the virtual reality symptom questionnaire (VRSQ) and Simulator sickness questionnaire (SSQ).
Opiod use peroperatively | Intraoperative (At the end of surgery)
  Rescue medication in case of block failure.
Patient satisfaction (7-point Likert scale) | Intraoperative (At the end of surgery)
  Patient satisfaction measured with the Patient Satisfaction Questionnaire and a 7-point Likert scale for measuring satisfaction rates with anesthesia, surgery and VR experience.
Needling time | Procedure (During performing the ultrasound-guided regional anesthesia block)
  The time from injection of the needle to the removal of the needle.
Surgical time | During surgery
  The time from incision to surgical completion

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nijs K, Treunen T, Jalil H, Lensen M, Wintmolders H, Keunen B, Vanloon M, Callebaut I, Geebelen L, Van de Velde M, Stessel B. Effect of virtual reality (VR) therapy on pain sensation in patients undergoing hand surgery under ultrasound-guided regional anesthesia: a randomized controlled trial. Reg Anesth Pain Med. 2025 Jun 1:rapm-2025-106418. doi: 10.1136/rapm-2025-106418. Online ahead of print. PMID 40451290